CLINICAL TRIAL: NCT07044765
Title: An Open-label, 2-arm, Single-sequence, Fed, Single Oral Dosing, Crossover Clinical Trial to Evaluate Safety and the Pharmacokinetics Between Dapagliflozin, Linagliptin and Metformin in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of Dapagliflozin, Linagliptin, and Metformin in Healthy Adults: Fed State Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AJU Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-IP013
Record Dates: First submitted 2025-06-17; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Two-period, single-dose, crossover study
  Interventions: Drug: Comparator 1; Drug: Comparator 2; Drug: Test Drug
- Group B (Experimental): Two-period, single-dose, crossover study (reversed order)
  Interventions: Drug: Comparator 1; Drug: Comparator 2; Drug: Test Drug

INTERVENTIONS:
Drug: Comparator 1 — Dapagliflozin 10mg + Linagliptin 5mg
Drug: Comparator 2 — Metformin 1000mg
Drug: Test Drug — Fixed-dose combination tablet (AJU-A53)

SUMMARY:
To Evaluate the Safety and Pharmacokinetics of Dapagliflozin, Linagliptin, and Metformin in Healthy Adults after taking the drugs with food (fed state).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged 19 to 50 years at the time of screening.
* Body mass index (BMI) between 18.0 and 30.0 kg/m², inclusive.

  * Male subjects must weigh ≥50 kg.
  * Female subjects must weigh ≥45 kg.
* No clinically significant congenital or chronic diseases requiring treatment, based on medical history and physical examination.
* Clinically acceptable results from laboratory tests (e.g., hematology, biochemistry, serology, urinalysis) and electrocardiogram (ECG) at screening, as determined by the investigator.
* Willing to use medically accepted contraception (excluding hormonal methods) from the first dose until 7 days after the last dose, and agrees not to donate sperm or eggs during this period.
* Able and willing to provide written informed consent after receiving a full explanation of the study.

Exclusion Criteria:

* Use of drugs known to induce or inhibit drug-metabolizing enzymes within 30 days prior to the first dose, or any medication likely to interfere with the study within 10 days prior to dosing.
* Participation in any clinical trial involving investigational products within 6 months prior to the first dose.
* Whole blood donation within 8 weeks, or component blood donation within 2 weeks prior to the first dose.
* History of gastrointestinal surgery that may affect drug absorption (excluding appendectomy and hernia repair).
* History of excessive alcohol consumption within 1 month prior to the first dose:

  * >21 drinks/week for males, >14 drinks/week for females (1 drink = 50 mL soju, 30 mL whiskey, or 250 mL beer)
* Known hypersensitivity to any component of the investigational product.
* Clinically significant renal, hepatic, cardiovascular, respiratory, metabolic, or infectious diseases, including but not limited to:

  * Moderate to severe renal impairment (eGFR or creatinine clearance <45 mL/min)
  * Dialysis
  * Acute or unstable heart failure
  * Acute myocardial infarction, septicemia, or shock
  * Type 1 diabetes, metabolic acidosis, or history of diabetic ketoacidosis
  * Major surgery planned during the study (except minor procedures not affecting food or fluid intake)
  * Severe infections, trauma, or nutritional deficiencies
* Positive pregnancy test or currently breastfeeding (for female subjects).
* History of significant psychiatric illness.
* Determined by the investigator to be unsuitable for the study for any other reason.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Cmax of Metformin | 0 hour ~ 48 hour after drug administration
  To assess the maximum observed plasma concentration (Cmax) of Metformin
AUCt of Metformin | 0 hour ~ 48 hour after drug administration
  To assess the plasma concentration-time curve from time 0 to the last measurable concentration (AUCt) of Metformin

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Gwangmyeong Hospital, Gwangmyeong, Gyeonggi-do, South Korea